CLINICAL TRIAL: NCT03597672
Title: A Prospective Cohort Study of Early Detection and Screening Strategy for Gatric Cancer in Sichuan Province China (SIGES-01)
Brief Title: Early Detection and Screening Strategy of Gatric Cancer in Sichuan Province-A Prospective Cohort Study (WCH-GC-SIGES-01)
Acronym: SIGES-01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jian-Kun Hu (Other)
Collaborators: Xin-Zu Chen (Unknown)
Responsible Party: Sponsor-Investigator, Jian-Kun Hu, Vice director of Gastrointestinal Surgery department, West China Hospital; Director of Institute of Gastric Cancer, State Key Laboratory of Biotherapy, West China Hospital, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: WCH-GC-SIGES-01; 320.2710.1815 (Other Grant/Funding Number: Wu Jieping Foundation's special fund for clinical research)
Record Dates: First submitted 2018-07-15; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Neoplasm, Stomach; H. Pylori Infection; Chronic Atrophic Gastritis
Keywords: Gastric carcinoma; Early diagnosis; screening stragety; health population cohort
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish prospective cohort of healthy population and corresponding serum sample bank in Sichuan province to provide platform for exploring early diagnosis and screening strategy of gastric cancer by a prospective cohort study.

DETAILED DESCRIPTION:
H. pylori was one of the most important carcinogenic factor for gastric cancer and play a crucial role in inducing gastritis, atrophy and canceration. Chronic atrophic gastritis (CAG) was a common precancerous disease, people with CAG become high-risk population and need regular follow-up. However, study about occurrence risk prediction for gastric cancer when H. pylori infection concurrence with CAG was still spare. In especial, there was still no population screening program based on serology. The relative clinical epidemiology for providing evidence for China gastric cancer screening program was very rare.

This study aim to evaluate gastric cancer occurrence risk and diagnostic value of people combined with H. pylori infection and CAG by Serological methods in Sichuan province China. We also project to design optimized screening program suitable for people in sichuan province China.

ELIGIBILITY:
Inclusion Criteria:

1. Inhabitant in Sichuan province in China (length of residence > 10 years);
2. Complete physical examination in our hospital, the outcomes was asymptomatic and cancer free healthy individuals;
3. Age between 20 and 70;
4. With normal cognitive and communication ability;
5. Without gastroscopy during recruitment, physical examination item including gastroscopy enrolled in prospective cohort study;
6. Wiling to accept 1-2 times routine physical examination in our hospital;
7. Agree to accept the follow-up of our project group;

Exclusion Criteria:

1. With history of malignant tumor;
2. Refuse to donate blood specimen;
3. With serious comorbidity and/or finite life (less than 5 years);
4. Request to retreat from this study;

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In our study, the poplatiion was enrolled among health inhabitant in Sichuan province in China. People who underwent physical examination in our center who statisfy our indications will be introdeced to participate in our study. The informed consent will be endosed and the blood sample will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of new cases of gastric carcinoma | 5 years
  The new cases of gastric and other epidermal malignant tumor

SECONDARY OUTCOMES:
Time of finding nee cases | 5 years
  The time during SIGES when finding nee gastric cancer and relative disease

CONTACTS AND LOCATIONS:
Locations (1):
- Jian-Kun Hu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
pending